CLINICAL TRIAL: NCT01957839
Title: Color Doppler Analysıs Of Uterin And Intraovarian Blood Flow Before And After Treatment Wıth Cabergoline In Hyperprolactinemic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Istanbul Bakirkoy Maternity and Children Diseases Hospital (Other Government)
Responsible Party: Principal Investigator, Osman Aşıcıoğlu, sisli etfal teaching hospital department gynecology and obstetric, Istanbul Bakirkoy Maternity and Children Diseases Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Aşıcıoğlu-08; OA8 (Other: Doppler)
Record Dates: First submitted 2013-09-10; First posted 2013-10-08 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: Adverse Reaction to Other Drugs and Medicines

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- pretreatment group (No Intervention): doppler evaluation at pretreatment period
- posttreatment group (Experimental): doppler evaluatıon in normoprolactinemia women who given cabergoline treatment
  Interventions: Drug: cabergoline treatment

INTERVENTIONS:
Drug: cabergoline treatment — cabergoline treatment for hyperprolactinemia group
  Arms: posttreatment group

SUMMARY:
the investigators examined the hypothesis that hyperprolactinemia may alter uterin, endometrial and intraovarian blood flow and may contribute to increased infertility by another way.

ELIGIBILITY:
Inclusion Criteria:

* Women who had blood prolactin level higher than 25ng/dl

Exclusion Criteria:

* Pregnancy
* Use of drugs effecting vasculature such as hormonal therapy, oral contraceptives, antihypertensives
* Diseases like pelvic inflammatory disease and systemic hypertension
* Women with clinically overt or treated cardiovascular disease
* Concurrent illness other than hyperprolactinemia

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2010-03; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
th effect of prolactin vascular flow and resistance | the effect of prolactin in vascular resistance at 2 weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Osman Temizkan, M.D., Principal Investigator — SİSLİ ETFAL TEACHİNG HOSPİTAL
Locations (1):
- Sisli Etfal Teaching Hosital, Şişli, Turkey (Türkiye)

REFERENCES:
- [Background] Ono M, Miki N, Amano K, Kawamata T, Seki T, Makino R, Takano K, Izumi S, Okada Y, Hori T. Individualized high-dose cabergoline therapy for hyperprolactinemic infertility in women with micro- and macroprolactinomas. J Clin Endocrinol Metab. 2010 Jun;95(6):2672-9. doi: 10.1210/jc.2009-2605. Epub 2010 Mar 31. PMID 20357175
- [Derived] Temizkan O, Temizkan S, Asicioglu O, Aydin K, Kucur S. Color Doppler analysis of uterine, spiral, and intraovarian artery blood flow before and after treatment with cabergoline in hyperprolactinemic patients. Gynecol Endocrinol. 2015 Jan;31(1):75-8. doi: 10.3109/09513590.2014.958989. Epub 2014 Sep 15. PMID 25222841